CLINICAL TRIAL: NCT04370808
Title: VITACOV: Vitamin D-related Polymorphisms and Vitamin D Levels as Risk Biomarkers of COVID-19 Infection Severity
Brief Title: VITACOV: Vitamin D Polymorphisms and Severity of COVID-19 Infection
Acronym: VITACOV
Status: Completed | Type: Observational
Sponsor: University of Lisbon (Other)
Collaborators: Cardiovascular Centre of Universidade de Lisboa (CCUL) (Unknown); Faculty of Medicine of Universidade de Lisboa (FMUL) (Unknown); Centro Hospitalar Universitário Lisboa Norte (Other); Centro Hospitalar Universitário São João (CHUSJ) (Unknown); CINTESIS - Center for Health Technology and Services Research (Unknown); Universidade Nova de Lisboa (Other); HeartGenetics, Genetics and Biotechnology SA (Industry); Instituto Gulbenkian de Ciência (IGC) (Unknown)
Responsible Party: Principal Investigator, Fausto J. Pinto, Professor, University of Lisbon
Other Study IDs: VITACOV
Record Dates: First submitted 2020-04-26; First posted 2020-05-01 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: COVID-19
Keywords: COVID-19; Vitamin D; Vitamin D polymorphisms
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mild to severe disease: Mild to severe disease (admission to isolation room)
  Interventions: Other: Exposure
- Critical patients: Critical patients (admission to ICU)
  Interventions: Other: Exposure

INTERVENTIONS:
Other: Exposure — Individuals with SARS-CoV-2 exposure and COVID-19 symptoms.

SUMMARY:
Vitamin D deficiency has been linked to hypertension, autoimmune, infectious and cardiovascular diseases which are risk factors for COVID-19. Moreover, COVID-19 patients have a very high prevalence of hypovitaminosis D (Turin data). Taken together, we aim to investigate whether genetic variants in vitamin D-related genes contribute to a poor COVID-19 outcome, particularly in hypertension and CV patients, proposing thus a personalized therapeutics based on vitamin D supplementation in order to reduce the severity and deaths.

DETAILED DESCRIPTION:
Collected data from Turin University indicate that hospitalized patients have a very high prevalence of hypovitaminosis D. Reports from China and Italy show that hypertension presents an increased risk of COVID-19-related death. Otherwise, observational studies suggest that 25(OH)D induces protection against respiratory pathogens while large-scale studies indicate that serum 25(OH)D-level is inversely correlated to hypertension prevalence. Recent published data (2020) shows that 66% of Portuguese adults present Vitamin D deficiency. HeartGenetics' genetic database with more than 8.500 Portuguese genotypes shows that the prevalence of vitamin D polymorphisms in this population is 4-fold higher than the EU average, increasing the risk of hypovitaminosis D.

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18 years and above.
* COVID-19 patients admitted with mild to severe disease (admission to isolation room) or critical patients (admission to ICU).
* Available to comply with study protocol and sign informed consent.

Exclusion Criteria:

* Patients diagnosed with COVID-19 not admitted to hospital.
* Patients unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-19 patients admitted to hospitals from Lisbon and Oporto.
Sampling Method: Non-Probability Sample
Enrollment: 517 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Differences in vitamin D blood levels between COVID-19 patients with different degrees of disease severity. | Blood samples of COVID-19 patients will be collected at baseline (after subject enrollment; single point collection).
Differences in genetic variants in vitamin D-related genes between COVID-19 patients with different degrees of disease severity. | Blood samples of COVID-19 patients will be collected at baseline (after subject enrollment; single point collection).

SECONDARY OUTCOMES:
Differences in vitamin D blood levels between COVID-19 patients in relation to mortality. | Through study completion, an average of 3 months.
Differences in vitamin D blood levels between COVID-19 patients in relation to length of stay in hospitals. | Through study completion, an average of 3 months.
Differences in vitamin D blood levels between COVID-19 patients in relation to duration of mechanical ventilation. | Through study completion, an average of 3 months.
Differences in genetic variants in vitamin D-related genes between COVID-19 patients in relation to mortality. | Through study completion, an average of 3 months.
Differences in genetic variants in vitamin D-related genes between COVID-19 patients in relation to length of stay in hospitals. | Through study completion, an average of 1 year.
Differences in genetic variants in vitamin D-related genes between COVID-19 patients in relation to duration of mechanical ventilation. | Through study completion, an average of 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Fausto J Pinto, PhD, Principal Investigator — Faculty of Medicine of Universidade de Lisboa; Conceição Calhau, PhD, Principal Investigator — Universidade Nova de Lisboa; Ana Freitas, PhD, Principal Investigator — HeartGenetics SA; Tiago Guimarães, PhD, Principal Investigator — Faculty of Medicine of the University of Porto; Ana Melo, PhD, Principal Investigator — BioData.pt/Instituto Gulbenkian Ciência
Locations (3):
- Portugal (3):
  - Cardiovascular Center at Universidade de Lisboa, Lisbon, Lisbon District
  - Centro Hospitalar Universitário Lisboa Norte, Lisbon, Lisbon District
  - Centro Hospitalar de São João, Porto

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Freitas AT, Calhau C, Antunes G, Araujo B, Bandeira M, Barreira S, Bazenga F, Braz S, Caldeira D, Santos SCR, Faria A, Faria D, Fraga M, Nogueira-Garcia B, Goncalves L, Kovalchuk P, Lacerda L, Lopes H, Luis D, Medeiros F, Melo AMP, Melo-Cristino J, Miranda A, Pereira C, Pinto AT, Pinto J, Proenca H, Ramos A, Rato JPR, Rocha F, Rocha JC, Moreira-Rosario A, Vazao H, Volovetska Y, Guimaraes JT, Pinto FJ. Vitamin D-related polymorphisms and vitamin D levels as risk biomarkers of COVID-19 disease severity. Sci Rep. 2021 Oct 21;11(1):20837. doi: 10.1038/s41598-021-99952-z. PMID 34675344